CLINICAL TRIAL: NCT05233904
Title: DART: Diagnostic-CT-Enabled Planning: A Randomized Trial in Palliative Radiation Therapy
Acronym: DART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, David Palma, Principle Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DART
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Advanced Cancer Requiring Palliative Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Patients will be booked for CT simulation and treatment as per the local institution's standard practice.
  Interventions: Diagnostic Test: Standard of Care
- Experimental Treatment Workflow (Experimental): Patients do not require a CT simulation appointment. A radiation treatment appointment will be scheduled on an optical surface guidance-equipped treatment unit as soon as available, but a minimum of 24 hours is required between EBAF processing and fraction 1.
  Interventions: Diagnostic Test: Diagnostic-CT-enabled Planning

INTERVENTIONS:
Diagnostic Test: Diagnostic-CT-enabled Planning — Diagnostic-CT-enabled planning for patient receiving palliative radiation treatment to bone, soft tissue and lung disease
  Arms: Experimental Treatment Workflow
Diagnostic Test: Standard of Care — Patients will be booked for CT simulation and treatment as per the local institution's standard practice
  Arms: Standard of Care

SUMMARY:
The objective of this trial is to assess the efficacy, acceptability, and scalability of diagnostic-CT-enabled planning, compared to conventional CT simulation planning.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to provide informed consent
* Patient has consented to PRT to bone/soft tissue metastases or primary targets in the thorax, abdomen, or pelvis and RO will use simple planning techniques (i.e. parallel-opposed pair or direct field beam arrangement)
* Patient will be scheduled for same-day simulation and treatment (if randomized to Arm 1)
* Patient has a pre-existing and recent (i.e. within 4 weeks of time of enrollment) diagnostic CT or CT-fused scan with full visualization of the region-of-interest which has been acquired from an approved diagnostic scanner
* Patient positioning scan is deemed acceptable and reproducible (e.g., patient is lying supine and relatively flat, there is no/minimal motion blur, ect.)
* Intravenous (IV)/oral contrast in the region-of-interest is permitted as long as it does not create artifact which obscured the target volume (density override calculations may be required)

Exclusion Criteria:

* Any contraindication to receiving radiation
* Oncologic emergencies and/or on-call cases
* Pregnant or lactating women
* Cases requiring composite dosimetric planning to account for previous radiotherapy or extended distance set-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Time in Centre (TIC) on Treatment Day | 1 Treatment Day
  This is defined as the total time in hours spent at the cancer centre from the scheduled CT simulation (Arrm 1) or treatment delivery (Arm 2) appointment until beam delivery completion.

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, MD, Principal Investigator — London Health Sciences Centre, Lawson Health Research Institute
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Neil M, Nguyen TK, Laba J, Dinniwell R, Warner A, Palma DA. DART: diagnostic-CT-enabled planning: a randomized trial in palliative radiation therapy (study protocol). BMC Palliat Care. 2022 Dec 9;21(1):220. doi: 10.1186/s12904-022-01115-y. PMID 36482335